CLINICAL TRIAL: NCT05105334
Title: Combined Treatment With Nonablative Fractional Laser and Radiofrequency Microneedling for the Treatment of Acne Scars: A Prospective, Randomized, Split-Face Study
Brief Title: Combined Therapy for Acne Scars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Goldman, Butterwick, Fitzpatrick and Groff (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Fraxel/Intracel-2021-8
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Atrophic Acne Scar
Keywords: Acne; Acne scar; Face; Microneedling; Intracel; Fraxel
MeSH Terms: conditions — Acne Vulgaris; Facies | interventions — Percutaneous Collagen Induction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, split-face, evaluator-blinded study
Who Masked: Outcomes Assessor
Masking Description: Clinical assessments and grading of severity of acne scarring will be performed by blinded-investigator assessment at each visit and at the post-treatment 3-month visit using live evaluations and photographs. At the 3-month follow up, three additional blinded dermatologists will clinically assess the severity of acne scarring.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nonablative fractional laser alone (Experimental)
  Interventions: Device: Nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alone
- Nonablative fractional laser alternating with microneedling with radiofrequency (Experimental)
  Interventions: Device: Nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alone; Device: Nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alternating with microneedling with radiofrequency (Intracel, Perigee Medical, Redwood City, CA)

INTERVENTIONS:
Device: Nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alone — Nonablative fractional 1550 nm erbium:glass laser. Settings: 40-70 mJ, treatment level 5-7 (14-20% coverage), 8 passes with cold air cooling (Zimmer MedizinSystems, Irvine, CA) set on level 5. To be repeated for a total of 4 sessions at 4-week intervals.
Device: Nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alternating with microneedling with radiofrequency (Intracel, Perigee Medical, Redwood City, CA) — Nonablative fractional 1550 nm erbium:glass laser. Settings: 40-70 mJ, treatment level 5-7 (14-20% coverage), 8 passes with cold air cooling (Zimmer MedizinSystems, Irvine, CA) set on level 5. This will be alternated with radiofrequency microneedling treatment will include 3 passes each at a depth of 2 mm, 1.5 mm, and 0.8 mm, treatment level 5 (32 w, 50 ms)-7 (40 w, 60 ms), monopolar setting with cold air cooling (Zimmer MedizinSystems, Irvine, CA) set on level 5. To be repeated for a total of 4 sessions (2 of each modality) at 4-week intervals.
  Arms: Nonablative fractional laser alternating with microneedling with radiofrequency

SUMMARY:
Compare the effectiveness of nonablative fractional resurfacing to radiofrequency micrnoeedling for facial acne scars in all skin types

DETAILED DESCRIPTION:
Quantify and compare the effectiveness of nonablative fractional laser (Fraxel re:store, Solta Medical, Bothell, WA) alone to nonablative fractional laser alternating with microneedling with radiofrequency (Intracel, Perigee Medical, Redwood City, CA) for the treatment of atrophic, facial acne scars in all skin types.

ELIGIBILITY:
1. Inclusion criteria

   1. Male or female in general good health ages 18 and older
   2. Fitzpatrick skin type I-VI
   3. Subject has completed an appropriately administered informed consent process which includes signing the IRB approved consent form
   4. Negative urine pregnancy test at baseline (if applicable)
   5. Willingness to have facial exams and digital photos performed of the face
   6. Moderate to severe atrophic acne scarring on the face per ECCA (échelle d'évaluation clinique des cicatrices d'acné) acne grading scale
   7. No change in estrogen releasing contraceptive method in 3 months, and no plans to change this contraceptive method during the course of the study
   8. No change in topical skin care
   9. Female patients will be either of non-childbearing potential defined as:

      1. Having no uterus
      2. No menses for at least 12 months. Or;

         Women of childbearing potential (WOCBP) must agree to use an effective method of birth control during the course of the study, such as:

      <!-- -->

      1. Oral contraceptive pill, injection, implant, patch, vaginal ring, intrauterine device
      2. Intrauterine coil
      3. Bilateral tubal ligation
      4. Barrier method used with an additional form of contraception (e.g., sponge, spermicide or condom)
      5. Abstinence (If practicing abstinence must agree to use barrier method described above (4) if becomes sexually active).
      6. Vasectomized partner (Must agree to use barrier method described above (4) if becomes sexually active with non-vasectomized).
2. Exclusion criteria

   1. Presence of incompletely healed wound in treatment area
   2. Pregnant, planning pregnancy or breastfeeding during the course of the study
   3. Energy-based device treatment in the treatment area in the last 6 months
   4. Treatments with a dermal filler or biostimulatory agent in the treatment area within the past 12 months
   5. Recent use of topical tretinoin, adapalene, tazarotene, hydroquinone, imiquimod, 5-fluorouracil, ingenol mebutate, concentrated hydrogen peroxide or diclofenac to the face within the previous 2 weeks.
   6. Individuals who have had a chemical peel or microdermabrasion of the face within 30 days prior to enrollment in the study
   7. Co-existing potentially confounding skin condition within treatment area (e.g. eczema, psoriasis, XP, rosacea) or the presence of suspected BCC or SCC in treatment area at investigator's discretion
   8. Has skin with open wounds, excessively sensitive skin, neurotic excoriations, dermatitis or inflammatory rosacea in the treatment area
   9. Individuals with known allergies or sensitivities to any of the ingredients of any topical products being used in this study (a list of the products with active and excipients will be provided below)
   10. Individuals with active psoriasis, eczema, sunburn, excessive scarring, tattoos, or other skin condition on the face that would interfere with the assessments of this study
   11. Subjects who participated on another study within the last 30 days
   12. Subjects currently on or planning to participate in any type of research study at another facility or a doctor's office during this study
   13. Subjects with a predisposition to keloid formation following surgery
   14. Subjects on systemic steroids (e.g. prednisone, dexamethasone), or topical steroids on the face which should be rigorously avoided prior to and throughout the course of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-11-08 (Estimated); Primary Completion 2022-05-08 (Estimated); Study Completion 2022-07-08 (Estimated)

PRIMARY OUTCOMES:
Change in atrophic acne scar | 3 months after final treatment
  The primary study endpoint will be clinical efficacy defined as change in atrophic acne scarring based on the ECCA grading scale and a 1-10 percentile scale.

SECONDARY OUTCOMES:
Subject comfort level | To be done right after treatments
  During each treatment visit patients will be asked to grade pain of treatment on a pain visual analog scale.
Subjective change | 3 months after final treatment
  Subjects will rate their perceived global change in acne scarring based on the subjected assessed global improvement scale.
Subject satisfaction | 3 months after final treatment
  Subjects will rate satisfaction on a 1-5 scale.
Adverse events | 3 months after final treatment
  To be recorded by treating physician after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Semsarzadeh, MD, Principal Investigator — Cosmetic Laser Dermatology

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan J, Kang S, Leyden J. Prevalence and Risk Factors of Acne Scarring Among Patients Consulting Dermatologists in the USA. J Drugs Dermatol. 2017 Feb 1;16(2):97-102. PMID 28300850
- [Background] Boen M, Jacob C. A Review and Update of Treatment Options Using the Acne Scar Classification System. Dermatol Surg. 2019 Mar;45(3):411-422. doi: 10.1097/DSS.0000000000001765. PMID 30856634
- [Background] Manstein D, Herron GS, Sink RK, Tanner H, Anderson RR. Fractional photothermolysis: a new concept for cutaneous remodeling using microscopic patterns of thermal injury. Lasers Surg Med. 2004;34(5):426-38. doi: 10.1002/lsm.20048. PMID 15216537
- [Background] Alster TS, Tanzi EL, Lazarus M. The use of fractional laser photothermolysis for the treatment of atrophic scars. Dermatol Surg. 2007 Mar;33(3):295-9. doi: 10.1111/j.1524-4725.2007.33059.x. PMID 17338686
- [Background] Hu S, Chen MC, Lee MC, Yang LC, Keoprasom N. Fractional resurfacing for the treatment of atrophic facial acne scars in asian skin. Dermatol Surg. 2009 May;35(5):826-32. doi: 10.1111/j.1524-4725.2009.01139.x. Epub 2009 Apr 6. PMID 19397671
- [Background] Hedelund L, Moreau KE, Beyer DM, Nymann P, Haedersdal M. Fractional nonablative 1,540-nm laser resurfacing of atrophic acne scars. A randomized controlled trial with blinded response evaluation. Lasers Med Sci. 2010 Sep;25(5):749-54. doi: 10.1007/s10103-010-0801-1. Epub 2010 Jun 17. PMID 20556471
- [Background] Bencini PL, Tourlaki A, Galimberti M, Longo C, Pellacani G, De Giorgi V, Guerriero G. Nonablative fractional photothermolysis for acne scars: clinical and in vivo microscopic documentation of treatment efficacy. Dermatol Ther. 2012 Sep-Oct;25(5):463-7. doi: 10.1111/j.1529-8019.2012.01478.x. PMID 23046026
- [Background] Al-Dhalimi M, Jaber A. Treatment of atrophic facial acne scars with fractional Er:Yag laser. J Cosmet Laser Ther. 2015;17(4):184-8. doi: 10.3109/14764172.2015.1007067. Epub 2015 Feb 13. PMID 25588037
- [Background] Alexis AF, Coley MK, Nijhawan RI, Luke JD, Shah SK, Argobi YA, Nodzenski M, Veledar E, Alam M. Nonablative Fractional Laser Resurfacing for Acne Scarring in Patients With Fitzpatrick Skin Phototypes IV-VI. Dermatol Surg. 2016 Mar;42(3):392-402. doi: 10.1097/DSS.0000000000000640. PMID 26945321
- [Background] Gold MH, Biron JA. Treatment of acne scars by fractional bipolar radiofrequency energy. J Cosmet Laser Ther. 2012 Aug;14(4):172-8. doi: 10.3109/14764172.2012.687824. Epub 2012 May 30. PMID 22548644
- [Background] Cho SI, Chung BY, Choi MG, Baek JH, Cho HJ, Park CW, Lee CH, Kim HO. Evaluation of the clinical efficacy of fractional radiofrequency microneedle treatment in acne scars and large facial pores. Dermatol Surg. 2012 Jul;38(7 Pt 1):1017-24. doi: 10.1111/j.1524-4725.2012.02402.x. Epub 2012 Apr 9. PMID 22487513
- [Background] Chandrashekar BS, Sriram R, Mysore R, Bhaskar S, Shetty A. Evaluation of microneedling fractional radiofrequency device for treatment of acne scars. J Cutan Aesthet Surg. 2014 Apr;7(2):93-7. doi: 10.4103/0974-2077.138328. PMID 25136209
- [Background] Vejjabhinanta V, Wanitphakdeedecha R, Limtanyakul P, Manuskiatti W. The efficacy in treatment of facial atrophic acne scars in Asians with a fractional radiofrequency microneedle system. J Eur Acad Dermatol Venereol. 2014 Sep;28(9):1219-25. doi: 10.1111/jdv.12267. Epub 2013 Sep 24. PMID 25158223
- [Background] Kaminaka C, Uede M, Matsunaka H, Furukawa F, Yamamoto Y. Clinical studies of the treatment of facial atrophic acne scars and acne with a bipolar fractional radiofrequency system. J Dermatol. 2015 Jun;42(6):580-7. doi: 10.1111/1346-8138.12864. Epub 2015 Apr 9. PMID 25855397
- [Background] Bulbul Baskan E, Akin Belli A. Evaluation of the efficacy of microneedle fractional radiofrequency in Turkish patients with atrophic facial acne scars. J Cosmet Dermatol. 2019 Oct;18(5):1317-1321. doi: 10.1111/jocd.12812. Epub 2018 Nov 11. PMID 30417509
- [Background] Jacob CI, Dover JS, Kaminer MS. Acne scarring: a classification system and review of treatment options. J Am Acad Dermatol. 2001 Jul;45(1):109-17. doi: 10.1067/mjd.2001.113451. PMID 11423843
- [Background] Zaleski-Larsen LA, Fabi SG, McGraw T, Taylor M. Acne Scar Treatment: A Multimodality Approach Tailored to Scar Type. Dermatol Surg. 2016 May;42 Suppl 2:S139-49. doi: 10.1097/DSS.0000000000000746. PMID 27128240
- [Background] Rongsaard N, Rummaneethorn P. Comparison of a fractional bipolar radiofrequency device and a fractional erbium-doped glass 1,550-nm device for the treatment of atrophic acne scars: a randomized split-face clinical study. Dermatol Surg. 2014 Jan;40(1):14-21. doi: 10.1111/dsu.12372. Epub 2013 Nov 25. PMID 24267397
- [Background] Chae WS, Seong JY, Jung HN, Kong SH, Kim MH, Suh HS, Choi YS. Comparative study on efficacy and safety of 1550 nm Er:Glass fractional laser and fractional radiofrequency microneedle device for facial atrophic acne scar. J Cosmet Dermatol. 2015 Jun;14(2):100-6. doi: 10.1111/jocd.12139. Epub 2015 Mar 23. PMID 25810322
- [Background] Kwon HH, Park HY, Choi SC, Bae Y, Kang C, Jung JY, Park GH. Combined Fractional Treatment of Acne Scars Involving Non-ablative 1,550-nm Erbium-glass Laser and Micro-needling Radiofrequency: A 16-week Prospective, Randomized Split-face Study. Acta Derm Venereol. 2017 Aug 31;97(8):947-951. doi: 10.2340/00015555-2701. PMID 28512669